CLINICAL TRIAL: NCT01323192
Title: A Double-blind, Placebo-controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of JNS001 in Adults With Attention-Deficit/Hyperactivity Disorder at Doses of 18 mg, 36 mg, 54 mg, or 72 mg Per Day
Brief Title: An Efficacy and Safety Study for JNS001 in Adults With Attention-Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR017755; JNS001-JPN-A01 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-03-10; First posted 2011-03-25 (Estimated); Results first posted 2013-09-06 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-06

CONDITIONS: Attention-Deficit Hyperactivity Disorder
Keywords: Concerta; Adults; Attention-Deficit/Hyperactivity Disorder; ADHD; Methylphenidate hydrochloride
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JNS001 (Experimental)
  Interventions: Drug: JNS001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNS001 — Participants will receive JNS001 (18 mg, 36 mg, 54 mg or 72 mg per day) orally once daily for 8 weeks.
  Arms: JNS001
Drug: Placebo — Participants will receive matching placebo orally once daily for 8 weeks.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy of JNS001 titrated to daily doses of 18 to 72 mg in adults with attention-deficit hyperactivity disorder (ADHD) relative to placebo.

DETAILED DESCRIPTION:
This is a randomized (the study drug is assigned by chance), double-blind (DB, neither physician nor patient knows the name of the assigned drug), multicenter, placebo-controlled, parallel group (each group of patients will be treated at the same time), dose-titration study. This study consists of a screening period, a DB phase (titration period and efficacy assessment period), and post-study phase. The study includes a 1 to 2-week screening period for wash-out of prohibited drugs, and screening for eligibility. Eligible patients will be randomly assigned to receive JNS001 or placebo in a ratio of 1:1. The study also includes a 4-week titration period. Patients will be titrated from a starting dose of 18 mg/day or matching placebo for 7 days (+/- 2 days), and continue with a weekly (+/- 2 days) increment of 18 mg until an individualized dose is achieved. Once an individualized dose is achieved, patients will remain on that dose for the rest of the titration period as far as tolerable. Doses can be tapered down only once during the titration period in the study, and their dose cannot be up-titrated again for the rest of the period. The 4-week titration period will be followed by the 4-week efficacy assessment period. The post-study phase for collection of additional safety data will be scheduled for 1 week after a patient's final study treatment. The study drug will be administered with water once daily in the morning at doses of 18 mg, 36 mg, 54 mg, 72 mg per day or the matching placebo. The study treatment period is 8 weeks (titration period of 4 weeks and efficacy assessment period of 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the criteria of ADHD (predominantly inattentive type [314.00], predominantly hyperactive-impulsive type [314.01], and combined type [314.01]) of DSM-IV-TR both at present and in childhood, based on Conners' Adult ADHD Diagnostic Interview for DSM-IV (CAADID) at screening
* DSM-IV Total ADHD Symptoms scores (18 items) of CAARS-O: SV score of = 24 as determined by investigator or co-investigator at baseline
* Healthy on the basis of physical examination, medical history, vital signs, 12-lead ECG and clinical laboratory tests performed at screening
* Women of childbearing potential must have a negative urine pregnancy test at screening
* Patients (and their legally-acceptable representative if patients are 18 or 19 years of age) must have signed an informed consent form (ICF), indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Presence or history of co-morbid psychiatric diagnosis per DSM-IV-TR criteria of bipolar I disorder, schizophrenia, schizoaffective disorder, or severe obsessive compulsive disorders
* Presence of co-morbid psychiatric diagnosis per DSM-IV-TR criteria of pervasive developmental disorder (including autistic disorder or Asperger's disorder), suicidality, or any other diagnosis that in the judgment the investigator or co-investigator would exclude the patient from the study
* Presence of motor tics, history of Tourette's disorder, or family history of Tourette's disorder
* Known or suspected mental retardation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 284 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (30):
- Japan (30):
  - Chiba
  - Chigasaki
  - Chiyoda City
  - Fuchū
  - Fukuoka
  - Fukushima
  - Hamamatsu
  - Higashiosaka
  - Ichikawa
  - Iruma
  - Isehara
  - Kashihara
  - Kishiwada
  - Kobe
  - Kumamoto
  - Kurume
  - Matsuyama
  - Nagasaki
  - Nagoya
  - Nara
  - Neyagawa
  - Osaka
  - Saitama
  - Sakai
  - Sapporo
  - Setagaya City
  - Shibuya City
  - Takatsuki
  - Tokyo
  - Yokohama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 39 study sites in Japan.
Pre-assignment Details: 284 participants were randomly assigned and treated with JNS001 or placebo in this study. One participant in the placebo group was excluded from the full analysis set because no post-dose efficacy data was available.
Groups:
- JNS001: Participants received JNS001 (18 mg, 36 mg, 54 mg or 72 mg per day) orally once daily for 8 weeks.
- Placebo: Participants received matching placebo orally once daily for 8 weeks.
Period: Overall Study
Arm/Group | JNS001 | Placebo
Started | 143 | 141
Completed | 134 | 135
Not Completed | 9 | 6
Not completed — Adverse Event | 6 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Noncompliance with study medication | 0 | 3
Not completed — Nonmedical reasons | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | JNS001 | Placebo | Total
Number analyzed (Participants) | 143 | 141 | 284
Age, Customized [Number; unit: Participants]
  18-24 years of age | 24 | 19 | 43
  25-35 years of age | 60 | 65 | 125
  36-49 years of age | 55 | 51 | 106
  50-64 years of age | 4 | 6 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 73 | 145
  Male | 71 | 68 | 139
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 143 | 139 | 282
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) Total Attention Deficit-Hyperactivity Disorder (ADHD) Symptoms Scores of Conners' Adult ADHD Rating Scale - Observer Screening Version (CAARS-O: SV)
Description: CAARS-O: SV evaluates DSM-IV-oriented inattention, impulsivity and hyperactivity as well as measures of self-concept. The CAARS-O:SV comprises 30 items to measure symptoms for ADHD in adults. Each item is scored from 0 (not at all, never) to 3 (very much, very frequently) with higher scores corresponding to worse symptoms. The total score can range from 0 (best) to 90 (worst). Lower score indicates improvement in ADHD symptoms.
Time Frame: Baseline (Day 0) to Endpoint (Week 8)
Population: Full analysis set: All participants who received at least 1 dose of study medication; and had baseline and at least 1 post-dose efficacy assessment. One participant in the placebo group was excluded from the full analysis set because no post-dose efficacy data was available.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | JNS001 | Placebo
Number analyzed (Participants) | 143 | 140
Scores on a scale | -12.5 (9.27) | -7.9 (9.61)
Statistical Analysis 1: Comparison: JNS001 vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in least square means = -4.5, 95% CI 2-sided [-6.7 to -2.4], Standard Error of Mean 1.10 — LS mean of JNS001 minus LS mean of Placebo

2. Secondary Outcome: Mean Change From Baseline to Endpoint in the Conners' Adult ADHD Rating Scale - Observer Screening Version (CAARS-O: SV) Total Score Other Than Total Attention Deficit-Hyperactivity Disorder (ADHD) Symptoms Score
Description: CAARS-O: SV evaluates DSM-IV-oriented inattention, impulsivity and hyperactivity as well as measures of self-concept. The CAARS-O: SV comprises 30 items to measure symptoms for ADHD in adults. Each item is scored from 0 (not at all, never) to 3 (very much, very frequently) with higher scores corresponding to worse symptoms. The total score can range from 0 (best) to 90 (worst). Lower score indicates improvement in ADHD symptoms.
Time Frame: Baseline (Day 0) to Endpoint (Week 8)
Population: Full analysis set: All participants who received at least 1 dose of study medication; and had baseline and at least 1 post-dose efficacy assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | JNS001 | Placebo
Number analyzed (Participants) | 143 | 140
Scores on a scale | -19.5 (15.42) | -12.5 (15.87)
Statistical Analysis 1: Comparison: JNS001 vs Placebo; Test type: Superiority or Other; p = 0.0002, ANCOVA; Difference in least square means = -6.9, Standard Error of Mean 1.83 — LS mean of JNS001 minus LS mean of Placebo

3. Secondary Outcome: Change From Baseline to Endpoint in Clinical Global Impression - Severity (CGI-S) Scores
Description: The CGI-S rating scale is used to rate the severity of a patient's psychotic condition on a 7-point scale. It is rated as follows: 1=Normal, not at all ill, 2=Borderline mentally ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Among the most extremely ill. Higher scores indicate worsening.
Time Frame: Baseline (Day 0) to Endpoint (Week 8)
Population: as for outcome 1
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | JNS001 | Placebo
Number analyzed (Participants) | 143 | 140
Scores on a scale | -1.0 (16.45) [-5 to 1] | -1.0 (16.55) [-4 to 2]
Statistical Analysis 1: Comparison: JNS001 vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA

4. Secondary Outcome: Clinical Global Impression of Change (CGI-C) Scores
Description: The CGI-C is a assessment of change in global clinical status, defined as a sense of well-being and ability to function in daily activities. CGI-C scores range from 1 (very much improved) through to 7 (very much worse). Higher scores indicate worsening.
Time Frame: Endpoint (Week 8)
Population: as for outcome 1
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | JNS001 | Placebo
Number analyzed (Participants) | 143 | 140
Scores on a scale | 3 [1 to 6] | 3 [1 to 6]
Statistical Analysis 1: Comparison: JNS001 vs Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA

5. Secondary Outcome: Mean Change From Baseline to Endpoint in the Conners' Adult Attention Deficit-Hyperactivity Disorder (ADHD) Rating Scales-Self Report: Screening Version (CAARS-S:SV) Score
Description: CAARS-S:SV evaluates DSM-IV-oriented inattention, impulsivity and hyperactivity as well as measures of self-concept. The CAARS-S:SV comprises 30 items to measure symptoms for ADHD in adults. Each item is scored from 0 (not at all, never) to 3 (very much, very frequently) with higher scores corresponding to worse symptoms. The total score can range from 0 (best) to 90 (worst). Lower score indicates improvement in ADHD symptoms.
Time Frame: Baseline (Day 0) to Endpoint (Week 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | JNS001 | Placebo
Number analyzed (Participants) | 143 | 140
Scores on a scale | -18.0 (16.45) | -10.9 (16.55)
Statistical Analysis 1: Comparison: JNS001 vs Placebo; Test type: Superiority or Other; p = 0.0003, ANCOVA; Difference in least square means = -6.9, Standard Error of Mean 1.83 — LS mean of JNS001 minus LS mean of Placebo

6. Secondary Outcome: Mean Change From Baseline to Endpoint in Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) Total Scores
Description: Q-LES-Q-SF is a 16-item questionnaire in which each question is rated on a 5-point scale with scores ranging from "1 = very poor" to "5 = very good". The total raw score is calculated by summing up the scores for the 16 items. The raw total score is transformed into a percentage maximum possible score using the following formula:(raw total score -minimum score) / (maximum possible raw score -minimum score). The minimum raw score on the Q-LES-Q-SF is 16 (worst), and the maximum score is 80 (best). A higher score indicates a better quality of life.
Time Frame: Baseline (Day 0) to Endpoint (Week 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | JNS001 | Placebo
Number analyzed (Participants) | 143 | 140
Scores on a scale | 2.4 (14.00) [-5 to 1] | 0.8 (12.69) [-4 to 2]
Statistical Analysis 1: Comparison: JNS001 vs Placebo; Test type: Superiority or Other; p = 0.4041, ANCOVA

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | JNS001 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/143 | 0/141
Other Adverse Events (participants affected / at risk) | 117/143 | 76/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JNS001 (N=143) | Placebo (N=141)
Psychotic disorder (Psychiatric disorders) | 1 | 0
Pneumothorax spontaneous tension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JNS001 (N=143) | Placebo (N=141)
Nasopharyngitis (Infections and infestations) | 24 | 19
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 57 | 10
Insomnia (Psychiatric disorders) | 15 | 14
Anxiety (Psychiatric disorders) | 6 | 3
Headache (Nervous system disorders) | 12 | 9
Dizziness (Nervous system disorders) | 6 | 2
Somnolence (Nervous system disorders) | 0 | 3
Tremor (Nervous system disorders) | 3 | 0
Palpitations (Cardiac disorders) | 26 | 2
Tachycardia (Cardiac disorders) | 8 | 0
Hot flush (Vascular disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 21 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 6
Abdominal discomfort (Gastrointestinal disorders) | 7 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Thirst (General disorders) | 20 | 6
Pyrexia (General disorders) | 7 | 0
Malaise (General disorders) | 6 | 0
Chest discomfort (General disorders) | 4 | 0
Weight decreased (Investigations) | 10 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 2
Blood triglycerides increased (Investigations) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days